CLINICAL TRIAL: NCT04152993
Title: Responsive Neurostimulation for Post-Traumatic Stress Disorder
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jean-PhilippeLangevin, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNS107673A
Record Dates: First submitted 2019-10-26; First posted 2019-11-06 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RNS group (Experimental): This study consists in only one arm. In this arm, the patients will undergo the placement of the RNS implant and the subsequent RNS programming to optimize the PTSD symptoms.
  Interventions: Device: NeuroPace® RNS® System

INTERVENTIONS:
Device: NeuroPace® RNS® System — In this intervention, patients suffering from PTSD undergo a surgical procedure to implant the responsive neurostimulation device (RNS, NeuroPace). This procedure involves the placement of a depth lead bilaterally in the amygdala and hippocampus following a trans-occipital trajectory. The two leads are then connected to a pulse generator fixated to the skull. RNS is able to detect specific signals from the target and to respond with a programmed electrical stimulation. One month after the implantation of the system, the patients will undergo 3 tasks: a fear conditioning task, the international affective picture system and the subsequent memory recall paradigm. These tasks will yield electrophysiological biomarkers of arousal and re-experiencing. We will then program RNS to detect and respond to those biomarkers. The patients will be followed longitudinally for improvement and evidence of target engagement as seen on cerebral metabolism and global electroencephalography.

SUMMARY:
Post-traumatic stress disorder (PTSD) refractory to treatment is marked by failure of fear extinction and its biological substrate, amygdala reactivity to trauma reminders. Decades of research have clarified the neuronal mechanisms coordinating fear extinction and consolidation. Fear cells and extinction cells in the basolateral amygdala (BLA) alter their firing rate based on the nature of the stimulus and the influence from the medial prefrontal cortex (mPFC) and the ventral hippocampus (vHPC). Together, the BLA, mPFC, and the vHPC form an anxiety-processing network where the BLA links stimulus to emotion, the vHPC provides memory context, and the mPFC coordinates extinction or consolidation. Local field potential (LFP) recordings from the BLA have revealed specific signals that correspond to an enhanced fear state. Previous studies have shown that neuromodulation of the BLA can promote extinction in a rodent model and in a treatment-refractory PTSD patient. This action is likely carried by disrupting fear signals within the BLA; however, continuous neurostimulation may also disrupt normal function of the amygdala. The present application proposes to investigate the use of Responsive Neurostimulation (RNS, Neuropace) in six (6) veterans suffering from severe treatment-resistant PTSD. This dual-activity device will allow us to chronically record LFPs from the BLA under specific conditions such as fear conditioning, exposure to trauma reminders, and emotional memory encoding and retrieval. In addition, the neural activity will be captured during real-life symptoms of flashback and nightmares. These recordings will provide the specific electrophysiological biomarkers of hypervigilance and re-experiencing. The device will then be programmed to detect and treat these biomarkers with a pre-determined electrical pulse. The patients will be followed prospectively using psychological scales but also with functional neuroimaging and electroencephalograms. These modalities will be used to determine the extent of circuit engagement as a result of the therapy. By approaching PTSD from a fear processing mechanism perspective, our project will serve as a proof of concept for other circuit-based therapies in psychiatry. This proposal is a multi-departmental effort involving 11 investigators across 7 departments and requires a close collaboration between clinical and basic scientists. As a result, the findings underlying chronic recordings will bridge the basic science results from fear conditioning research to clinical neural processes in PTSD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 25-60 years.
2. Able to give informed consent in accordance with institutional policies and participate in the 4-year follow-up, involving assessments and stimulator adjustments.
3. Patients must be stable on their current psychotropic medication for a period of 2 months before implantation and agree to not increase dosages or add any new medications for the first 6 months of the study, unless medically necessary.
4. Chart diagnosis of chronic and treatment-refractory PTSD as the principal psychiatric diagnosis and cause of distress and social/occupational impairment.
5. Confirmation of PTSD as the primary psychiatric diagnosis by the study psychiatrist via clinical interview and CAPS.
6. Minimum 5-year total illness duration, with no 6-month period of clinical remission during the 2 years prior to entry in the study.
7. Stage 2 level of treatment resistance as per Sippel et al.136: Clinical record documented failure to respond to adequate (minimum 3 month, with adherence) trials of at least 3 of the following evidence-based treatments including at least one pharmacologic agent below, and at least one trauma-focused individual cognitive-behavior psychotherapy among the following: Pharmacologic: sertraline, paroxetine, fluoxetine or venlafaxine, at maximally tolerated FDA recommended doses. Psychotherapy: Prolonged Exposure Therapy (PE); Cognitive Processing Therapy (CPT); Eye movement Desensitization and Reprocessing (EMDR); or other form of evidence-based cognitive behavior therapy for PTSD
8. Patients who are unable to complete trauma-focused psychotherapy may be included if they began treatment, and the cause of treatment cessation was that the risks of further treatment, including intense psychological suffering, outweighed the potential benefits of continuing the treatment.
9. All evidence-based psychotherapy for PTSD has been completed a minimum of 3 months prior to enrolment.
10. Minimum baseline past month CAPS-5 Score of 47, with full PTSD diagnostic criteria met, and scores of ≥ 3 on at least one item from the intrusive (CAPS-5 items 1-5) and hyperarousal (CAPS-5 Items 15-20) clusters; and this severity maintained for at least one month during the baseline period based on two separate measures.
11. Clinically significant impairment in occupational functioning due to PTSD, manifested by one or more of the following: a) Total federal (service connected ≥ 70%), or State (SSI) disability compensation for at least the past 2 years for PTSD; b) global assessment of functioning score ≤ 45; c) no period of full time gainful employment ≥ 3 months in the past 5 years. Or clinically significant impairment in social functioning due to PTSD, manifested by one or more of the following: (i) little or no social activity outside the household other than as necessary for medical appointments, practical matters such as grocery shopping, or to interact with other veterans; (ii) reliable description by a spouse or significant other, living with the patient, of repeated avoidance/refusal to participate in customary social engagements with friends, family or for recreational activities due to PTSD; (iii) two or more verbal or physical interpersonal altercations within the past year requiring another person's intervention to prevent further escalation, or involving law enforcement.
12. Presence in the veteran's life of a spouse, family member or friend who can confirm the symptoms and impairment from PTSD and lack of symptomatic remission in the past 2 years; participate with the study psychiatrist in answering questions about symptoms and functioning at scheduled follow-up visits; and report unexpected adverse neurological or psychiatric events to study investigators and, if advised by study investigators, assist the patient in accessing necessary services to address obtain care.
13. Willingness to have unexpected neurological or psychiatric symptom shared with the study psychiatrists and other study clinicians.
14. Other medical conditions must be stable for at least 1 year, (conditions that require intermittent use of steroids or chemotherapy are excluded).

Exclusion Criteria:

1. Suicide attempt in the last 2 years and/or presence of a suicide plan (an answer of "Yes" to Question C4 in Section C-Suicidality of MINI International Neuropsychiatric Interview);
2. Unstable psychosis or bipolar disorder; significant acute or ongoing risk for violence;
3. Patients primarily diagnosed with DSM-IV-TR Axis I disorder other than PTSD as determined by the MINI;
4. Within the 3 months prior to enrolment, subject has started a new psychotherapy program;
5. Alcohol or illicit substance use disorder within the last 6 months, unstable remission of substance abuse, or chart evidence that co-morbid substance use disorder could account for lack of treatment response;
6. Current significant neurological conditions, including epilepsy, stroke, movement disorder; history of serious head injury with loss of consciousness if associated with neurological or neuropsychological deficit that could interfere with study participation or outcome assessment; or if associated with structural MRI abnormality.
7. Uncontrolled medical condition including cardiovascular problems and diabetes;
8. Uncontrolled chronic pain;
9. Baseline Montgomery Asberg Depression Rating Scale (MADRS) of ≥ 28;
10. Use of warfarin;
11. Significant abnormality on preoperative structural brain MRI;
12. ECT in the past 6 months;
13. Contraindications to MRIs or the need for recurrent body MRIs;
14. Immunosuppression;
15. High risk for surgery;
16. Current pursuit of new or increased disability compensation for PTSD;
17. Intracranial implants (aneurysm clip, shunt, cochlear implant, electrodes);
18. Patient has had past cranial neurosurgery;
19. Use of other investigational drugs within 30 days of baseline.
20. Patients suffering from a neurovascular condition or other intracranial process.
21. Patients suffering from a condition associated with a significant cognitive impairment.

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Spectral power analysis and oscillatory properties | Baseline
  This is associated with Specific Aim 1: To determine electrophysiological biomarkers of fear, extinction and PTSD symptoms. The metric for measurement will be Better Oscillation Detection (BOSC)
Spectral power analysis and oscillatory properties | through study completion, an average of 1 year
  This is associated with Specific Aim 1: To determine electrophysiological biomarkers of fear, extinction and PTSD symptoms. The metric for measurement will be Better Oscillation Detection (BOSC)
Cross-frequency coupling and power coherence comodulograms | Baseline
  This is associated with Specific Aim 1: To determine electrophysiological biomarkers of fear, extinction and PTSD symptoms. The metric for measurement will be modulation index.
Cross-frequency coupling and power coherence comodulograms | through study completion, an average of 1 year
  This is associated with Specific Aim 1: To determine electrophysiological biomarkers of fear, extinction and PTSD symptoms. The metric for measurement will be modulation index.
Region of Interest analysis (FDG PET) | Baseline
  This is associated with Specific Aim 2: To determine engagement of fear processing neural networks by neurostimulation. The metric for measurement will be Cerebral metabolic rate of glucose (CMRglc)
Region of Interest analysis (FDG PET) | After initial exposure session
  This is associated with Specific Aim 2: To determine engagement of fear processing neural networks by neurostimulation. The metric for measurement will be Cerebral metabolic rate of glucose (CMRglc)
Region of Interest analysis (FDG PET) | 12 months post-operatively
  This is associated with Specific Aim 2: To determine engagement of fear processing neural networks by neurostimulation. The metric for measurement will be Cerebral metabolic rate of glucose (CMRglc)
Alpha rhythm frequency (EEG) | Baseline
  This is associated with Specific Aim 2: To determine engagement of fear processing neural networks by neurostimulation. The metric for measurement will be frequency (Hertz)
Alpha rhythm frequency (EEG) | monthly after implantation for the first year
  This is associated with Specific Aim 2: To determine engagement of fear processing neural networks by neurostimulation. The metric for measurement will be frequency (Hertz)
Alpha rhythm frequency (EEG) | quarterly during year 2-4
  This is associated with Specific Aim 2: To determine engagement of fear processing neural networks by neurostimulation. The metric for measurement will be frequency (Hertz)
Source localization (EEG) | Baseline
  This is associated with Specific Aim 2: To determine engagement of fear processing neural networks by neurostimulation. The metric for measurement will be discrete dipole fitting.
Source localization (EEG) | through study completion, an average of 1 year
  This is associated with Specific Aim 2: To determine engagement of fear processing neural networks by neurostimulation. The metric for measurement will be discrete dipole fitting.

SECONDARY OUTCOMES:
Clinician Administered PTSD Scale | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score.
Clinician Administered PTSD Scale | monthly after implantation for the first year
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score.
Occurrence of adverse events | through study completion, an average of 1 year
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by frequency/severity.
Psychological scales (HAMA) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Psychological scales (HAMA) | monthly after implantation for the first year
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Psychological scales (HAMA) | every three months up to 48 months after baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Psychological scales (MADRS) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Psychological scales (MADRS) | monthly after implantation for the first year
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Psychological scales (MADRS) | every three months up to 48 months after baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Psychological scales (YBOC) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Psychological scales (YBOC) | monthly after implantation for the first year
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Psychological scales (YBOC) | every three months up to 48 months after baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Digit Span subtest | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Digit Span subtest | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Trail Making Test A and B | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Trail Making Test A and B | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Ruff Figural Fluency Test (RFFT) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Ruff Figural Fluency Test (RFFT) | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Brief Visual Memory Test | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Brief Visual Memory Test | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Revised (BVMT-R) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Revised (BVMT-R) | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
California Verbal Learning Test | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
California Verbal Learning Test | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Attention, Processing Speed and Memory: Wechsler Adult Intelligence Scale IV (WAIS-IV)143 - Digit Span subtest, Trail Making Test A and B, Ruff Figural Fluency Test (RFFT), Brief Visual Memory Test - Revised (BVMT-R), California Verbal Learning Test | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Attention, Processing Speed and Memory: Wechsler Adult Intelligence Scale IV (WAIS-IV)143 - Digit Span subtest, Trail Making Test A and B, Ruff Figural Fluency Test (RFFT), Brief Visual Memory Test - Revised (BVMT-R), California Verbal Learning Test | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Wechsler Adult Intelligence Scale IV (WAIS-IV) | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Wechsler Adult Intelligence Scale IV (WAIS-IV) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Wechsler Test of Adult Reading | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Wechsler Test of Adult Reading | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Controlled Oral Word Association (COWAT) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Controlled Oral Word Association (COWAT) | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Hooper Visual Organization Test (VOT) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Hooper Visual Organization Test (VOT) | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Rey-Osterrieth Complex Figure Test (CFT) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Rey-Osterrieth Complex Figure Test (CFT) | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Wisconsin Card Sorting Test (WCST) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Wisconsin Card Sorting Test (WCST) | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Stroop Color and Word Test | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Stroop Color and Word Test | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Iowa Gambling Task (IGT) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Iowa Gambling Task (IGT) | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Montreal Cognitive Assessment (MOCA) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Montreal Cognitive Assessment (MOCA) | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Frontal Systems/ Executive Functions: Wisconsin Card Sorting Test (WCST), Stroop Color and Word Test, Iowa Gambling Task (IGT) | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Rey-15 Recognition test of Mental Effort | Months 6, 12, 24 and 48
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
Rey-15 Recognition test of Mental Effort | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
SF-36V (quality of life) | Baseline
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score
SF-36V (quality of life) | through study completion, an average of 1 year
  This is associated with Specific Aim 3: To assess the efficacy and safety of BLA stimulation for treatment-resistant PTSD. This test will be measured by the score

CONTACTS AND LOCATIONS:
Locations (1):
- VA Greater Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The data obtained will be shared semi-annually. The data shared will include de-identified raw scores on the assessments, PET study analysis and safety data (adverse events, EEG findings). We will insure the accuracy of the data being shared and we will work with the NCDT staff in order to confirm that we are submitting the data appropriately.
  We will also comply with the NIH Public Access Policy during any publication related to this study.
Supporting Information: CSR
Time Frame: The data will become available on a semiannual basis.

REFERENCES:
- [Derived] Gill JL, Schneiders JA, Stangl M, Aghajan ZM, Vallejo M, Hiller S, Topalovic U, Inman CS, Villaroman D, Bari A, Adhikari A, Rao VR, Fanselow MS, Craske MG, Krahl SE, Chen JWY, Vick M, Hasulak NR, Kao JC, Koek RJ, Suthana N, Langevin JP. A pilot study of closed-loop neuromodulation for treatment-resistant post-traumatic stress disorder. Nat Commun. 2023 May 24;14(1):2997. doi: 10.1038/s41467-023-38712-1. PMID 37225710